CLINICAL TRIAL: NCT01073774
Title: Side by Side - Prediction of Couples' Adjustment to Breast or Gynecological Cancer
Acronym: Side by Side
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universitaet Braunschweig (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: DFG, DFG
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: He61491994; DFG He61481994
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Enhancing Couples Coping
Keywords: breast cancer couples coping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Side by Side (Experimental)
  Interventions: Behavioral: Side by side
- couples control condition (Active Comparator)
  Interventions: Behavioral: couples control condition

INTERVENTIONS:
Behavioral: Side by side
  Arms: Side by Side
Behavioral: couples control condition
  Arms: couples control condition

SUMMARY:
The diagnosis and treatment of cancer leads to emotional distress, and major disruptions in role functioning. Traditionally, psychosocial services offer individuals diagnosed with cancer peer group support or individual counseling with only few consideration of type or stage of cancer. Besides most cancers significantly impacting not only the individual but also their partners and families, breast and gynecological cancer may be particularly embedded in an interpersonal context, namely in the couple's relationship. Breast and gynecological cancer cause additional concerns about the women' body image, sexual functioning and these cancers may be prone to provoke or enhance maladaptive patterns of interaction between women and their partners. Thus, not only the individual but also the couple's functioning is threatened by these diagnoses.

The aim of the here proposed study is to identify predictors of couple's adjustment and to help couples to improve their ability to support each other during this time. In a multi-site study, we will evaluate the efficacy of a couple-based intervention entitled "Side by Side: Coping with Cancer Together ("Seite an Seite: Krebs Gemeinsam Bewältigen"). The intervention teaches couples relationship skills that have been repeatedly validated within the marital field. The aim of the intervention is to improve couples' skills to talk to each other effectively about cancer-related topics, and enhance (or maintain) an affectionate relationship in the face of death.

We will randomly assign 303 women recently diagnosed with either breast or gynecological cancer and their partners to one of two conditions: (1) Seite an Seite, or (2) Treatment-As-Usual, in which couples receive no active psychosocial intervention. Assessment will be conducted pre-, post-, and at 6 and 12 months follow-up. These assessments include for both partners negative and positive self-report measures of individual functioning (such as mood, anxiety and benefit finding) and relationship functioning (such as relationship distress, communication patterns). Furthermore, at pre-, post- and 12-month Follow-up observational data on mutual supportive behavior when communicating about a cancer-related topic will be collected. The study may enhance our understanding of the significance of relationship skills in the process of adjusting to cancer as a couple and as an individual.

ELIGIBILITY:
Inclusion Criteria:

* woman was recently diagnosed with breast cancer (Stage I - III)
* no history of other cancers
* woman and her male partner were married or have been living in a committed relationship for at least 12 month
* both partners are willing to participate and able to speak German

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)